CLINICAL TRIAL: NCT05980052
Title: Goal Setting to Promote Physical Activity Adherence in Midlife to Reduce Risk of Alzheimer's Disease and Related-Dementias: A Randomized Mechanistic Proof-Of-Concept Trial
Brief Title: Goal Setting to Promote Physical Activity Adherence in Midlife Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00016394; R61AG078089 (NIH)
Record Dates: First submitted 2023-07-17; First posted 2023-08-07 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Physical Activity; Exercise
Keywords: exercise; physical activity; mild cognitive impairment; Alzheimer's disease; dementia; behavior change; midlife
MeSH Terms: conditions — Motor Activity; Cognitive Dysfunction; Alzheimer Disease; Dementia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Four arm randomized mechanistic proof-of-concept trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Static weekly physical activity goal of 150 minutes/week (Experimental): Participants will receive a physical activity action planning intervention and assigned a static weekly physical activity goal of 150 minutes/week of moderate-intensity activity; action planning sessions will focus on the participant achieving this weekly goal.
  Interventions: Behavioral: Physical Activity
- Incremental weekly physical activity goal increase (Experimental): Participants will receive a physical activity action planning intervention and assigned a weekly physical activity goal that is 20% greater than the level of moderate-intensity physical activity performed the previous week; action planning sessions will focus on the participant achieving their assigned goal.
  Interventions: Behavioral: Physical Activity
- Self-selected weekly physical activity goal (Experimental): Participants will receive a physical activity action planning intervention and will self-select their own moderate-intensity physical activity goal each week; action planning sessions will focus on helping participants achieve their self-selected goal.
  Interventions: Behavioral: Physical Activity
- No stated weekly physical activity goal (comparison group) (Experimental): Participants will receive a physical activity action planning intervention that does not include explicitly stated physical activity goals to achieve.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Theory-driven behavioral physical activity promotion intervention.

SUMMARY:
Engaging in regular physical activity during midlife is a key lifestyle behavior associated with reduced risk for Alzheimer's disease and related dementias (AD/ADRD). Yet nearly half of midlife adults (48%) do not meet national physical activity guidelines. The purpose of this mechanistic trial is to identify effective goal setting techniques to enhance psychosocial processes of self-regulation for the successful promotion of PA and adherence to national PA guidelines among midlife adults, with the long-term goal of reducing AD/ADRD risk

DETAILED DESCRIPTION:
More than 6 million U.S. adults live with diagnoses of Alzheimer's Disease and Related Dementias (AD/ADRD), with projections as high as 13.8 million cases by 2050. There are no cures for AD/ADRD, making lifestyle factors key targets for reducing risk, as they account for at least a third of AD/ADRD cases. Engaging in regular physical activity (PA), particularly in midlife, is associated with reduced risk for AD/ADRD. Yet, nearly half of midlife adults (48%) do not meet national PA guidelines of 150 minutes/week of moderate-intensity PA. Goal setting is a commonly used behavior change strategy to increase PA. Key psychosocial mechanisms believed to underpin the use of goal setting to promote PA include self-regulation and self-efficacy. However, the most effective goal setting technique to enhance these psychosocial mechanisms for the successful promotion of PA and adherence to national PA guidelines remains unclear. In the proposed study, the investigators will use a two-phased approach to empirically test three goal setting techniques to enhance psychosocial mechanisms of self-regulation and self-efficacy for the successful promotion of PA and adherence to national PA guidelines among insufficiently active midlife adults with obesity. In the R61 phase, a Phase 1 pilot study will establish feasibility and help refine the intervention. In the R33 phase, a Phase 2 9-month 4-arm proof-of-concept mechanistic trial (6-month active intervention and 3-month no contact follow-up) will be implemented to establish preliminary efficacy of goal setting techniques to increase PA and promote adherence to national PA guidelines. All participants will receive a Fitbit to self-monitor PA and engage in PA action planning sessions with a study interventionist. In addition, participants will be randomly assigned to 1 of 4 groups: i) static weekly goal of 150 minutes/week of moderate-intensity PA, which most closely resembles the approach of public health campaigns and care providers; ii) weekly self-selected PA goals, which allows for self-determination and adaptation of the goal; iii) modest incremental weekly PA increase goal (i.e., researcher determined PA goal that 20% minutes/week greater than the minutes/week of PA in the previous week); or iv) non-goal setting control group. Based on Goal Setting Theory, it is hypothesized that participants in the incremental goal group will have the greatest increases in self-regulation and self-efficacy, which in turn, will lead to the greatest improvements in PA and adherence to national PA guidelines over the 9-month intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45 to 65 years
* BMI between 30 kg/m2 to 50 kg/m2
* Participants must weigh a minimum of 110 pounds
* Engaging in 60 minutes or less of self-reported moderate-to-vigorous physical activity at screening (based on Exercise Vital Sign Questionnaire)
* Self-reported ownership of a smartphone with an iOS or Android operating system (necessary for participants to track their activity using a Fitbit activity monitor)

Exclusion Criteria:

* Endorsing an item on the Physical Activity Readiness Questionnaire (PAR-Q), unless a physician's note is provided
* Resting blood pressure greater than 200/110 mmHG as assessed at the baseline study assessment (unless a physician's note is provided)
* Pregnant or planning to become pregnant in next 8-months (Phase 1) or 12 months (Phase 2)
* Plans to relocate out of metropolitan Phoenix, Arizona area in the next 8-months (Phase 1) or 12 months (Phase 2)
* Participation in another physical activity, nutrition or weight loss program at time of screening or at any time during the intervention
* Individuals with mild cognitive impairment (MCI), as determined by either a self-report of receiving a diagnosis of MCI from a health care provider or as assessed by the Montreal Cognitive Assessment (MoCA) at the study orientation session. A score < 26 is an exclusion criterion for US born participants. A score of <23 is an exclusion for participants born outside of the US who completed their high school education in a country where English is not the primary language.
* Being previously prescribed one of the 5 approved Alzheimer's medications, including: Donepezil (Aricept), Rivastigmine (Exelon), Galantamine (Razadyne), Memantine (Namenda), Memantine + Donepezil (Namzaric)
* Score of 16 or higher on the Center for Epidemiological Studies-Depression Scale (CES-D)
* Self-reported current diagnosis of major depression
* Currently taking 2 or more ant-depression drugs
* History of stroke
* Incarcerated individuals (i.e., Prisoners)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in accelerometer-measured moderate-to-vigorous intensity physical activity from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Participants will wear wrist-worn ActiGraph GT9X Link Activity monitors the activity monitor on their non-dominant wrist during all waking hours for 7 consecutive days to provide an assessment of usual activity.
Change in Fitbit-assessed moderate-to-vigorous intensity physical activity | Assessed daily up to 9-months
  Participants will wear a wrist-worn Fitbit activity monitor daily throughout the 9-month intervention.
Change in self-reported moderate-to-vigorous intensity physical activity from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Self-reported minutes per week of moderate-to-vigorous physical activity assessed by the 7-day Physical Activity Recall.

SECONDARY OUTCOMES:
Change in physical activity self-regulation from baseline to 6- and 9-months | Assessed monthly up to 9-months
  Assessed using the The 12-item Physical Activity Self-Regulation Scale (PASR-12; Umstattd et al., 2009). This scale assess 6 PA-related self-regulatory domains: self-monitoring, goal setting, eliciting social support, reinforcements, time management, relapse prevention. The range of possible scores is 5-60, with higher scores indicating higher levels of physical activity self-regulation.
Change in physical activity behavioral strategies from baseline to 6- and 9-months | Assessed monthly up to 9-months
  Assessed using 10-item Self-Regulation scale from the Health Belief Survey (Anderson et al., 2010) This scale assesses the use of behavioral strategies to incorporate physical activity into daily activities (i.e., take stairs instead of elevator, walking instead of driving when running errands). The range of possible scores for this measure is 1-5, with higher scores indicating higher levels of physical activity self-regulation.
Change in physical activity self-efficacy from baseline to 6- and 9-months | Assessed monthly up to 9-months
  Assessed by the 12-item Exercise Self-Efficacy survey (Sallis et al.1987). The range of possible scores for this measure is 1-5, with higher scores indicating higher levels of physical activity self-efficacy.
Change in general self-regulation from baseline to 6- and 9-months | Assessed monthly up to 9-months
  Assessed using the 31-item short version of the self-regulation scale (SSRS; Carey, Neal, & Collins, 2004). The range of possible scores is 31 to 155, with higher scores indicate greater self-regulation
Change in General Self-Efficacy from baseline to 6- and 9-months | Assessed monthly up to 9-months
  Assessed using the 10-item Self-Efficacy Scale publicly available in SOBC repository & NIH Toolbox. The range of possible scores is 31 to 155. Higher scores indicate greater self-efficacy.

OTHER OUTCOMES:
Change in immediate verbal memory from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Assessed using the Auditory Verbal Learning Test. This test is administered on an iPad and is scored automatically using software available from the NIH Toolbox, which provides an age-adjusted standard score (possible range: 50 to 150) and percentile score (possible range: 1st percentile to 99th percentile). Higher scores indicate greater immediate verbal memory capacity.
Change in delayed verbal memory from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Assessed using the Delayed Auditory Verbal Learning Test. This test is administered on an iPad and is scored automatically using software available from the NIH Toolbox, which provides an age-adjusted standard score (possible range: 50 to 150) and percentile score (possible range: 1st percentile to 99th percentile). Higher scores indicate greater immediate verbal memory capacity.
Change in visual memory from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Assessed using the Picture Sequence Memory Test. This test is administered on an iPad and is scored automatically using software available from the NIH Toolbox, which provides an age-adjusted standard score (possible range: 50 to 150) and percentile score (possible range: 1st percentile to 99th percentile). Higher scores indicate greater immediate verbal memory capacity.
Change in executive function from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Assessed using the Dimensional Change Card Sort Test. This test is administered on an iPad and is scored automatically using software available from the NIH Toolbox, which provides an age-adjusted standard score (possible range: 50 to 150) and percentile score (possible range: 1st percentile to 99th percentile). Higher scores indicate greater immediate verbal memory capacity.
Change in pattern comparison processing speed from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Assessed using the Pattern Comparison Processing Speed Test. This test asks participants to determine whether two stimuli are the same or not the same as quickly as possible without making mistakes. It is administered on an iPad and is scored automatically using software available from the NIH Toolbox, which provides an age-adjusted standard score (possible range: 50 to 150) and percentile score (possible range: 1st percentile to 99th percentile). Higher scores indicate greater immediate verbal memory capacity.
Change in processing speed from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Assessed using the Oral Symbol Digit Test. This test assesses time needed to process pairings of digits & symbols and is administered on an iPad and is scored automatically using software available from the NIH Toolbox, which provides an age-adjusted standard score (possible range: 50 to 150) and percentile score (possible range: 1st percentile to 99th percentile). Higher scores indicate greater immediate verbal memory capacity.
Change in plasma amyloid 42/40 ratio from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Assessed using commercial Meso Scale Discovery (MSD) assays
Change in plasma phosphorylated tau 231 from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Assessed using commercial Meso Scale Discovery (MSD) assays
Adjudication for Mild Cognitive Impairment (MCI) | Performed using data collected at 6-months and 9-months
  Investigator-consensus adjudication will be performed by three investigators to determine if a participant has diagnosable MCI according to the NIA-AA guidelines (Albert et al., 20211).
Change in body weight from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Measured in kilograms using an electronic scale
Change in BMI from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Calculated using the formula: weight (in kilograms) / height (in meters)^squared
Change in blood pressure (mmHG) from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Both systolic and diastolic blood pressure will be assessed using electronic sphygmomanometer following 5-min rest
Change in fasting plasma glucose (mg/dL) from baseline to 6- and 9-months | baseline, 6-months, 9-months
  Assessed using an automated chemistry analyzer
Change in serum lipids (mg/DL) from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Triglycerides, total cholesterol, LDL-C, and HDL-C will be assessed
Change in insulin sensitivity (µIU/mL) from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Calculated using homeostatic model assessment (HOMA)
Change in depressive symptoms from baseline to 6- and 9-months | Assessed at baseline, 6-months, 9-months
  Assessed using the 20-item Center for Epidemiologic Studies Depression Scale (CES-D; Radloff, 1977). This scale has a possible score range 0 to 60, with higher scores indicating greater frequency of depressive symptoms.
Protocol Adherence | Assessed at 6-months and 9-months
  Number of days Fitbit worn, number of days Fitbit synced, number of weeks study arm specific PA goal met, and number of individual coaching meetings attended.
Treatment acceptance | Assessed at 6-months and 9-months
  Survey assessing acceptance, feasibility, and consumer satisfaction of intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided